CLINICAL TRIAL: NCT06033391
Title: Promoting Mental Health in Adolescents Through Mobile Apps: the Case of Obsessive-compulsive Disorder
Brief Title: Mobile App for Obsessive-compulsive Disorder in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, Gemma García-Soriano, PhD, associate professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2557724
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Obsessive-Compulsive Disorder in Adolescence
Keywords: obsessive-compulsive disorder; cognitive therapy; maladaptive beliefs; mobile app; adolescence
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Participants that meet the inclusion criteria will complete the web-based baseline assessment (pre), with questionnaires relating to maladaptive beliefs, mood (anxiety and depressions), self-esteem and OCD symptoms. After, experimental group will use the GGOC-AD, and control group will use the GGN-AD for 14 days. Then, both groups will complete again the above-mentioned assessment instruments (post use of the app). Finally, all participants will complete the follow-up measures at one month.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GGOC-AD (GG Obsessive-Compulsive Disorder - Adolescents) (Experimental): The experimental group will use the GGOC-AD module for 14 days after the first assessment.
  Interventions: Device: GGOC-AD (GG Obsessive-Compulsive Disorder - Adolescents)
- GGN-AD (GG Neutral - Adolescents) (Active Comparator): The control group will use the GGN-AD module for 14 days after the first assessment.
  Interventions: Device: GGN-AD (GG Neutral - Adolescents)

INTERVENTIONS:
Device: GGOC-AD (GG Obsessive-Compulsive Disorder - Adolescents) — GGOC was originally designed to challenge maladaptive beliefs that underline OCD symptoms in adult population. It was adapted to adolescent population. It consists of statements that are presented to the user, and that can portray either negative ("I can't trust myself") or positive beliefs ("I have a lot of good characteristics"). Users have to respond by either pulling these towards "Accept" or "Reject".
  Arms: GGOC-AD (GG Obsessive-Compulsive Disorder - Adolescents)
Device: GGN-AD (GG Neutral - Adolescents) — it was designed to have a comparison group. It consists of neutral statements such as "Madrid is a Spanish city", that ought not to produce changes in the direction of our hypothesis. These have to be "Accepted" or "Rejected" based on their veracity.
  Arms: GGN-AD (GG Neutral - Adolescents)

SUMMARY:
The aim of the present study is to assess the efficacy of the module GGOC-AD (GG Obsessive-Compulsive Disorder - Adolescents) in reducing obsessive-compulsive disorder (OCD) related maladaptive beliefs and OCD symptoms in adolescents from 15 to 18 years old. Specifically, a randomized controlled trial with two conditions (experimental and control) will be carried out in a non-clinical adolescent population to assess pre-post-intervention changes. After 14 days of using GGOC-AD, it is expected, primarily, to find a decrease in OCD-related maladaptive beliefs and OCD symptoms. As secondary results, we do not expect changes in emotional symptomatology, but we do expect an increase in self-esteem. Additionally, these changes are expected to be found in a one-month follow-up.

DETAILED DESCRIPTION:
Pediatric OCD is a serious problem and, if not treated early on, is associated with significant impairment. The app GGOC, aimed at working on OCD-related dysfunctional beliefs in adults, has proven in previous studies in adult clinical and non-clinical samples, to significantly decrease maladaptive beliefs associated with OCD and obsessive-compulsive symptomatology. Also, it can significantly increase self-esteem. Therefore, it is relevant to adapt the GGOC application to the adolescent population (GGOC-AD) and evaluate its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. To have signed the informed consent, both the adolescents and their parents or legal guardians.
2. Being enrolled in 4th level of Obligatory Secondary Education of the Spanish Education System (ISCED levels 2 and 3 in the International Standard Classification of Education)
3. To have a mobile phone (indistinctly Android or iOS mobile system) with Internet access.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Change in obsessive beliefs | Through app completion (14 days) and 1 month follow-up
  Score change in obsessive compulsive maladaptive beliefs measured by the Obsessive Beliefs Questionnaire-Child Version (OBQ-CV). Total score is computed as a mean of the 44 items, ranging from 0 "strongly disagree" to 4 "strongly agree". Higher scores indicate the person has more obsessive beliefs.
Change in obsessive-compulsive symptomatology | Through app completion (14 days) and 1 month follow-up
  Score change in obsessive-compulsive symptoms measured by the Obsessive Compulsive Inventory- Child Version (OCI-R-CV). Total score is computed as a mean of the 21 items, ranging from 0 "never" to 2 "always". Higher scores indicate a greater presence of obsessive-compulsive symptoms.

SECONDARY OUTCOMES:
Change in emotional symptoms | Through app completion (14 days) and 1 month follow-up
  Change in depression and anxiety symptoms measured by The Patient Health Questionnaire for Depression and Anxiety (PH-4). It consists of 4 items, two for Anxiety and two for Depression, with a 4-point Likert scale (from 0 = "never" to 3 = "almost every day"). Higher scores indicate a greater presence of depression or anxiety symptoms.
Change in self-esteem | Through app completion (14 days) and 1 month follow-up
  Change in score of Single Item Self Esteem Scale (SISE). Self-Esteem is measured with this single item ranging from 1 "It is not very true for me" to 7 "It is very true for me". Higher scores indicate a higher self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma García-Soriano, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia/ Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Share all IPD that underlie results in a publication.
Time Frame: It will be available after the publication of the study.
Access Criteria: Data will be available in a repository website: Zenodo.
URL: https://zenodo.org/

REFERENCES:
- [Background] Roncero M, Belloch A, Doron G. Can Brief, Daily Training Using a Mobile App Help Change Maladaptive Beliefs? Crossover Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Feb 13;7(2):e11443. doi: 10.2196/11443. PMID 30758294
- [Derived] Saman Y, Pascual-Vera B, Corberan M, Arnaez S, Roncero M, Garcia-Soriano G. A mobile app to challenge obsessional beliefs in adolescents: a protocol of a two-armed, parallel randomized controlled trial. BMC Psychiatry. 2024 Apr 9;24(1):265. doi: 10.1186/s12888-024-05735-x. PMID 38594680
- See also: Link to download the app from Google Play — https://play.google.com/store/apps/details?id=air.com.samuramu.gg.oc